CLINICAL TRIAL: NCT04448275
Title: Effect of Neurodynamics Nerve Flossing on Femoral Neuropathy in Haemophilic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T./REC /012/002733
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Femoral Neuropathy in Haemophilic Patients
Keywords: Neurodynamics,; Nerve flossing;; femoral neuropathy; , haemophilia,
MeSH Terms: conditions — Femoral Neuropathy; Hemophilia A

STUDY DESIGN:
Intervention Model Description: control group which received conventional selected exercise program in form of Ultrasound therapy The flexibility exercises for iliopsoas & quadriceps The iliopsoas & quadriceps muscles strength exercise
  and study group received the same exercise training program in addition to Neurodynamics Nerve flossing three times per week for three successive months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received conventional selected exercise program and in addition to Neurodynamics Nerve flossing for femoral nerve
  Interventions: Other: Neurodynamics Nerve flossing; Other: conventional selected exercise program
- control group (Experimental): received conventional selected exercise program in form of: Ultrasound therapy The flexibility exercises for iliopsoas & quadriceps in heamophilic patient The iliopsoas & quadriceps muscles strength exercise
  Interventions: Other: conventional selected exercise program

INTERVENTIONS:
Other: Neurodynamics Nerve flossing — Neurodynamics Nerve flossing for femoral nerve that includes two techniques inform of:
  "slider technique" and the second is the "tensioner technique
  Arms: study group
Other: conventional selected exercise program — Ultrasound therapy The flexibility exercises for iliopsoas & quadriceps The iliopsoas & quadriceps muscles strength exercise

SUMMARY:
To investigate the effect of Neurodynamics Nerve flossing on femoral neuropathy in patients with haemophilia

Background: heamophilia is one of the serious chronic disorders in children and adolescents which results in less physical activities and restlessness hours than their peer.

HYPOTHESES:

This study will hypnotize that:

Neurodynamics Nerve flossing will have a significant effect on femoral neuropathy in patients with haemophilia

RESEARCH QUESTION:

will the Neurodynamics Nerve flossing has an effect on femoral neuropathy in patients with haemophilia?

DETAILED DESCRIPTION:
Haemophilic patients with Femoral Neuropathy will be randomly divided in two equal groups control group which will receive conventional selected exercise program and study group will receive the same exercise training program in addition to Neurodynamics Nerve flossing three times per week for three successive months.

The Evaluation will done pre and post interventions included:

femoral nerve motor conduction velocity, muscle test For Iliopsoas and Quadriceps muscles and Pain visual analogue scale.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia A or B, all the patients
* positive femoral nerve tension test
* the Manual muscle test for iliopsoas and quadriceps muscles in all patients not less than grade 2 according to the oxford scale
* the age ranging from (12:16) years
* all the participants will be able to communicate verbally ,obey commands and instructions and co-operate with testing and training protocols

Exclusion Criteria:

* any participants have auditory, visual and sever cardiac disorders
* Patients who have mild degree of hemophilia
* Patients who have joint, muscle bleeding or pain in the lower limb in the preceding 3 weeks
* patients with any other neurological disorders or musculoskeletal disorders or deformities of the lower limb.

Ages: 12 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Electromyography Nerve conduction study | 12 weeks
  Femoral Nerve motor conduction velocity (m/sec.) , via the Neuropack S1 MEB9004 EMG device
Femoral Nerve Tension Test, for femoral nerve injury | 12 weeks
  Femoral Nerve Tension Test is a neural tension test used to stress the femoral nerve
  A positive test was be reproduction of the patient's symptoms as burning discomfort in the groin or anterior thigh occurred if there was femoral nerve involvement.
Manual muscle test, Oxford five grades of muscle power assessment | 12 weeks
  The group Manual muscle test was used for testing the strength of iliopsoas and quadriceps muscles, according to the Oxford Scale as the Muscle strength is often rated on a scale of 0/5 as follow:
  (0/5) no contraction of muscle, (1/5) muscle flicker contraction, but no movement (2/5) movement possible, but not against gravity (test the joint in its horizontal plane), (3/5) movement possible against gravity, but not against resistance by the therapist, (4/5) movement possible against some resistance by the examiner and (5/5) normal strength

CONTACTS AND LOCATIONS:
Overall Officials: Lama S Mahmoud, PHD, Study Director — lecturer , department of Neuromuscular Disorders and its surgery, faculty of physical therapy O6U physical therapy
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No